CLINICAL TRIAL: NCT00006119
Title: Phase II Study of Hydroxyurea for the Treatment of Recurrent and/or Nonoperable Meningioma
Brief Title: Hydroxyurea in Treating Patients With Recurrent and/or Unresectable Meningioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068132; FRE-FNCLCC-98009; EU-20018
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult grade III meningioma; adult grade I meningioma; adult grade II meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Meningioma | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: hydroxyurea

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of hydroxyurea in treating patients who have recurrent and/or unresectable meningioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine complete, partial, or stable response to hydroxyurea in patients with recurrent and/or nonresectable meningioma.
* Determine response at 2 years to this regimen in these patients.
* Determine overall and disease free survival of these patients after this regimen.
* Determine quality of life of these patients.
* Determine the toxicities of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to grade of disease (I vs II or III).

Patients receive oral hydroxyurea daily for 2 years.

Quality of life is assessed before treatment, then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 60 patients (30 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven progressive meningioma that is not curable by surgery

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Over 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST and ALT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN

Renal:

* Creatinine no greater than 2 times ULN

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after study
* No other malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent corticosteroids allowed for control of intracranial pressure

Radiotherapy:

* Prior radiotherapy allowed
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 1 year since prior experimental therapy

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-07 (Actual); Primary Completion 2004-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Frappaz, MD, Study Chair — Centre Leon Berard
Locations (5):
- France (5):
  - Hopital Saint Andre, Bordeaux
  - Centre Leon Berard, Lyon
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours